CLINICAL TRIAL: NCT06707688
Title: Abbott Medical - VERITAS Study
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10523; G240218 (Other: FDA IDE Number)
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation (AF); Stoke
Keywords: Left Atrial Appendage; LAA Occluder; Afib; Amulet; Abbott; VERITAS
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Amulet™ 2 Left Atrial Appendage (LAA) Occluder (Experimental): Transcatheter left atrial appendage (LAA) occluder
  Interventions: Device: Amulet™ 2 Left Atrial Appendage (LAA) Occluder

INTERVENTIONS:
Device: Amulet™ 2 Left Atrial Appendage (LAA) Occluder — Patient will undergo the implantation of the Amulet™ 2 Left Atrial Appendage (LAA) Occluder

SUMMARY:
The primary objective of this study is to evaluate the safety and effectiveness of Abbott's Amulet™ 2 Left Atrial Appendage (LAA) occluder device (Amulet 2 device) in patients who have non-valvular atrial fibrillation and who are at increased risk for stroke and systemic embolism and have appropriate rationale to seek a non-pharmacologic alternative to oral anticoagulation.

ELIGIBILITY:
Inclusion Criteria:

1. Paroxysmal, persistent, permanent or long-term/longstanding persistent non-valvular AF and has not been diagnosed with rheumatic mitral valve disease
2. CHA2DS2-VASc score of ≥2 for males or ≥3 for females
3. Has an appropriate rationale to seek a non-pharmacologic alternative to oral anticoagulation
4. Subject is eligible to stop anticoagulation if the LAA is sealed based on the implanting physician's opinion
5. Subject is able to comply with the protocol defined pharmacologic regimen following Amulet 2 device implant (as described in Section 6.5)
6. Subject is able to understand and willing to provide written informed consent to participate in the clinical investigation
7. Subject is able and willing to return for required follow-up visits and protocol required clinical investigation activities
8. 18 years of age or older, or the age of legal consent

Exclusion Criteria:

1. Required to take P2Y12 platelet inhibitor beyond 6 months when Amulet 2 LAA Occluder implant procedure would occur
2. Is considered at high risk for general anesthesia in the opinion of the Investigator or based on past adverse reaction(s) requiring medical intervention or which resulted in prolongation of hospital stay
3. Atrial septal defect or patent foramen ovale repair or occluder
4. Implanted with a mechanical valve prosthesis
5. Subject anatomy will not accommodate or is contraindicated for transesophageal echocardiography probe use (e.g., presence of esophageal varices, esophageal stricture, or history of esophageal cancer), or subject has experienced adverse events related to transesophageal echocardiography acquisition or has refused transesophageal echocardiography acquisition in the past
6. Underwent any cardiac or non-cardiac intervention or surgery within 30 days prior to when Amulet 2 device implant procedure would occur (any intervention or surgery that utilized anesthesia, anesthetic, or sedation)
7. Underwent catheter ablation for AF or atrial flutter within 60 days prior to when Amulet 2 device implant procedure would occur
8. Inpatient hospitalization due to clinical event or other sequelae within the past 7 days (i.e., not related to planned clinical study procedure or assessments)
9. Subject is planning any cardiac or non-cardiac intervention or surgery within 60 days after when Amulet 2 device implant procedure would occur (any intervention or surgery that utilized anesthesia, anesthetic, or sedation), except for study related activities
10. Inferior vena cava filter present
11. Left ventricular ejection fraction ≤30% (per most recent assessment)
12. Experienced stroke or transient ischemic attack within 90 days prior to when Amulet 2 device implant procedure would occur
13. Experienced myocardial infarction (with or without intervention) within 90 days prior to when Amulet 2 device implant procedure would occur
14. New York Heart Association (NYHA) Class IV Congestive Heart Failure
15. Known symptomatic carotid disease (defined as > 50% lumen diameter narrowing on CTA, MRA, or TCD with symptoms of ipsilateral transient or visual TIA evidenced by amaurosis fugax, ipsilateral hemispheric TIAs or ipsilateral stroke); if subject has a history of carotid stent or endarterectomy the subject is eligible if there is < 50% lumen diameter narrowing
16. Underwent prior attempted endocardial, epicardial, or surgical LAA closure or occlusion, defined as deployment of a device or surgical procedure whether successful or unsuccessful
17. Reversible cause of AF (i.e., secondary to thyroid disorders, acute alcohol intoxication, trauma, recent major surgical procedures)
18. History of idiopathic or recurrent venous thromboembolism within the past 5 years
19. Thrombocytopenia (defined as < 50,000 platelets per microliter (<50 x 109/L) or anemia (defined as hemoglobin < 10 g/dL) requiring transfusions
20. Known hypersensitivity to any portion of the device material or individual components of the Amulet 2 device (e.g., nickel allergy)
21. Actively enrolled in, or plans to enroll in, a concurrent clinical investigation in which the active treatment arm may confound the results of the VERITAS Study. Each instance must be brought to the attention of the Sponsor to determine eligibility.
22. Is pregnant or breastfeeding, or pregnancy is planned during the course of the investigation
23. Active endocarditis or other infection producing bacteremia
24. Transient case of AF (i.e., never previously detected, provoked/induced by surgical or catheter manipulations, etc.)
25. Severe renal failure (estimated glomerular filtration rate <30 ml/min/1.73m2) or on chronic dialysis
26. Life expectancy is less than 2 years in the opinion of the Investigator
27. Presence of other anatomic or comorbid conditions, or other medical, social, or psychological conditions that, in the Investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow up requirements, or impact the scientific soundness of the clinical investigation results.

Anatomical Exclusion Criteria:

1. Intracardiac thrombus
2. Existing circumferential pericardial effusion >2 mm
3. Mitral valve stenosis, defined as a mitral valve area of <1.5 cm2
4. Inter-atrial communication (PFO/ASD with right to left shunt, if TEE performed) with an atrial septal aneurysm (excursion >15 mm or length ≥15 mm; excursion defined as maximal protrusion of the atrial septal aneurysm beyond the plane of the atrial septum) or large shunt (i.e., during Valsalva maneuver ≥20 bubbles of right-to-left shunt within 3 cardiac cycles after contrast media enters the right atrium, if TEE performed)
5. Complex atheroma of the descending aorta and/or aortic arch, defined as plaque >4 mm in thickness, plaque ulceration, and/or mobile lesions
6. Cardiac tumor
7. LAA anatomy that cannot accommodate the Amulet 2 device, as per manufacturer's IFU (i.e., the LAA size must be within the sizing chart of the Amulet 2 device)
8. Placement of the device would damage or interfere with the function of any intracardiac or intravascular structure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 458 (Actual)
Dates: Start 2024-11-11 (Actual); Primary Completion 2025-11-04 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
The primary safety endpoint is the occurrence of any prespecified safety events through 7 days post-procedure or hospital discharge, whichever is later. | 7 days post-procedure or hospital discharge
  The primary safety endpoint is the occurrence of any of the following events through 7 days post-procedure or hospital discharge, whichever is later: death, ischemic stroke, systemic embolism, or device/procedure related complications requiring open cardiac surgery or major endovascular intervention. Device/procedure related events contributing to the primary endpoint may include pseudoaneurysm or AV fistula repair, whereas percutaneous drainage of pericardial effusion, snaring of embolized devices, thrombin injection or nonsurgical treatment of access site complications will not contribute to the primary endpoint.
The primary effectiveness endpoint is LAA occlusion defined as no peri-device flow or peri-device flow ≤5mm based on TEE/TOE at the 45-day follow-up visit. | 45 days
  The primary effectiveness endpoint is LAA occlusion defined as no peri-device flow or peri-device flow ≤5mm based on Doppler color flow TEE/TOE at the 45-day follow-up visit as assessed by an independent core laboratory.

SECONDARY OUTCOMES:
The secondary effectiveness endpoint is the composite of ischemic stroke or systemic embolism at 24 months. | 24 months
  The secondary effectiveness endpoint is the composite of ischemic stroke or systemic embolism at 24 months.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan Palmer, Study Director — Abbott Medical; Devi Nair, MD, Principal Investigator — Arrhythmia Research Group; Mohamad Alkhouli, MD, Principal Investigator — Mayo Clinic
Locations (35):
- United States (19):
  - Arizona Arrhythmia Research Group, Phoenix, Arizona
  - Arrhythmia Research Group, Jonesboro, Arkansas
  - Baptist Medical Center, Jacksonville, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Northside Hospital, Atlanta, Georgia
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - Henry Ford Providence Southfield Hospital, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - CHI Health Creighton University Medical Center-Bergan Mercy, Omaha, Nebraska
  - NYU Langone Health, New York, New York
  - Mount Sinai Hospital, New York, New York
  - Roper Hospital, Charleston, South Carolina
  - Trident Medical Center, Charleston, South Carolina
  - Vanderbilt Heart & Vascular Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Baylor Scott & White All Saints Medical Center, Fort Worth, Texas
  - Vital Heart and Vein, Humble, Texas
  - Baylor Scott & White - The Heart Hospital Plano, Plano, Texas
  - Heart Rhythm Associates, Shenandoah, Texas
- Hôpital Civil Marie Curie, Lodelinsart, Belgium
- Canada (2):
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - Institut de Cardiologie de Montreal (Montreal Heart Inst.), Montreal, Quebec
- Denmark (2):
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen
- France (2):
  - CHU Gabriel Montpied, Clermont-Ferrand, Auvergn
  - Institute Cardio. Paris-Sud - Institut Jacques Cartier, Massy
- Germany (4):
  - Cardioangiologisches Centrum am Bethanien Krankenhaus, Frankfurt am Main, Hesse
  - Deutsches Herzzentrum der Charité, Berlin
  - Universitätsklinikum Schleswig-Holstein - Campus Lübeck, Lübeck
  - Heinrich-Braun-Klinikum gemeinnützige gGmbH Standort Zwickau, Zwickau
- Ospedale San Raffaele, Milan, Italy
- Spain (3):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario de Salamanca, Salamanca
- Center Inselspital Bern, Bern, Canton of Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No